CLINICAL TRIAL: NCT00531206
Title: Observational Non-interventional Study About Antiretroviral Combination Treatment With Aptivus in Combination With Low-dose Ritonavir in HIV Type 1 Infected Patients
Brief Title: Observational Non-interventional Study (Anwendungsbeobachtung) With Aptivus® (Tipranavir) in HIV-infected Patients.
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 1182.112
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Results first posted 2010-05-12 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- All participants
  Interventions: Drug: Tipranavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Tipranavir
Drug: Ritonavir — low dose

SUMMARY:
This observational study is supposed to assess (under conditions of clinical practice in daily routine) whether treatment with Aptivus (tipranavir) in combination with low-dose Norvir (ritonavir) will durably suppress viral load and may achieve suppression of viral load below the limit of detection.

ELIGIBILITY:
Inclusion Criteria:

Highly pre-treated male and female adult patients with virus resistant to multiple protease inhibitors. Aptivus (tipranavir), co-administered with low dose Norvir (ritonavir), is indicated for combination antiretroviral treatment of HIV-1 infection in highly pre-treated adult patients with virus resistant to multiple protease inhibitors.

Exclusion Criteria:

* Age < 18 years
* pregnant female patients
* Hypersensitivity to the active substance or to any of the excipients.
* Patients with moderate or severe (Child-Pugh B or C) hepatic impairment.
* Rifampicin should not be used with Aptivus (tipranavir) because co-administration may cause large decreases in tipranavir concentrations which may in turn significantly decrease the tipranavir therapeutic effect.
* Herbal preparations containing St John's wort must not be used while taking Aptivus (tipranavir) due to the risk of decreased plasma concentrations and reduced clinical effects of tipranavir.
* Co-administration of Aptivus (tipranavir) with low dose Norvir (ritonavir), with active substances that are highly dependent on CYP3A for clearance and for which elevated plasma concentrations are associated with serious and/or life-threatening events is contraindicated. These active substances include antiarrhythmics (amiodarone, bepridil, quinidine), antihistamines (astemizole, terfenadine), ergot derivatives (dihydroergotamine, ergonovine, ergotamine, methylergonovine), gastrointestinal motility agents (cisapride), neuroleptics (pimozide, sertindole), sedatives/hypnotics (triazolam) and HMG-CoA reductase inhibitors (simvastatin and lovastatin). In addition, co-administration of Aptivus (tipranavir) with low dose Norvir (ritonavir), with drugs that are highly dependent on CYP2D6 for clearance, such as the antiarrhythmics flecainide and propafenone, is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2006-08; Primary Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (27):
- Germany (27):
  - Boehringer Ingelheim Investigational Site, Aachen
  - Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site, Bremen
  - Boehringer Ingelheim Investigational Site, Cologne
  - Boehringer Ingelheim Investigational Site, Dortmund
  - Boehringer Ingelheim Investigational Site, Düsseldorf
  - Boehringer Ingelheim Investigational Site, Erlangen
  - Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site, Giessen
  - Boehringer Ingelheim Investigational Site, Halle
  - Boehringer Ingelheim Investigational Site, Hamburg
  - Boehringer Ingelheim Investigational Site, Hanover
  - Boehringer Ingelheim Investigational Site, Homburg/Saar
  - Boehringer Ingelheim Investigational Site, Karlsruhe
  - Boehringer Ingelheim Investigational Site, Krefeld
  - Boehringer Ingelheim Investigational Site, Leipzig
  - Boehringer Ingelheim Investigational Site, Magdeburg
  - Boehringer Ingelheim Investigational Site, Mainz
  - Boehringer Ingelheim Investigational Site, München
  - Boehringer Ingelheim Investigational Site, Münster
  - Boehringer Ingelheim Investigational Site, Nuremberg
  - Boehringer Ingelheim Investigational Site, Oldenburg
  - Boehringer Ingelheim Investigational Site, Osnabrück
  - Boehringer Ingelheim Investigational Site, Saarbrücken
  - Boehringer Ingelheim Investigational Site, Stuttgart
  - Boehringer Ingelheim Investigational Site, Wuppertal

RESULTS

PARTICIPANT FLOW:
Groups:
- Aptivus® in Combination With Low-dose Norvir®: Aptivus® in combination with low-dose Norvir® and optimised backbone therapy
Period: Overall Study
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Started | 65
Completed | 45
Not Completed | 20
Not completed — Adverse Event related | 5
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 5
Not completed — including non-related adverse events | 8

BASELINE CHARACTERISTICS:
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 59

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: The safety and tolerability of the observed antiretroviral therapy were based on the Adverse Events (AEs) and Serious Adverse Events (SAEs) reported in the case report forms.
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Number; unit: Number of patients with adverse events
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
Number of patients with adverse events | 23

2. Secondary Outcome: Change in Viral Load
Description: Log10 change from baseline in viral load over time
Time Frame: Baseline and 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Median (Inter-Quartile Range); unit: log10 copies/ml
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
log10 copies/ml
  change from baseline to month 1 (4 weeks) | -1.56 [-1.94 to -0.54]
  change from baseline to month 3 (12 weeks) | -1.70 [-2.47 to -0.48]
  change from baseline to month 6 (24 weeks) | -1.42 [-2.59 to -0.45]
  change from baseline to month 9 (36 weeks) | -1.42 [-2.94 to -0.71]
  change from baseline to month 12 (52 weeks) | -1.45 [-2.42 to -0.54]

3. Secondary Outcome: CD4+ Cell Count
Description: Change from baseline in CD4+ count over time
Time Frame: Baseline and 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
cells/mm3
  change from baseline to month 1 (4 weeks) | 30.50 [-17.0 to 85.5]
  change from baseline to month 3 (12 weeks) | 43.50 [-4.5 to 144.5]
  change from baseline to month 6 (24 weeks) | 39.50 [0.0 to 144.0]
  change from baseline to month 9 (36 weeks) | 63.00 [13.0 to 155.0]
  change from baseline to month 12 (52 weeks) | 36.00 [-5.0 to 191.0]

4. Secondary Outcome: Subjective Well-being
Description: Investigator's opinion of patient's general condition (quality of life)
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Number; unit: participants
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
participants
  good general condition | 23
  moderate general condition | 35
  bad general condition | 7
  missing | 0

5. Secondary Outcome: Serious Adverse Events
Description: as for outcome 1
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Number; unit: Number of patients
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
Number of patients | 3

6. Secondary Outcome: Deaths
Description: as for outcome 1
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Number; unit: Number of patients
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
Number of patients | 1

7. Secondary Outcome: Discontinuations Due to an Adverse Event
Description: as for outcome 1
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Number; unit: Number of patients
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
Number of patients | 6

8. Secondary Outcome: Adverse Events Related to Therapy With Tipranavir/Ritonavir Based on Investigator's Opinion
Description: as for outcome 1
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Number; unit: Number of patients
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
Number of patients | 7

9. Secondary Outcome: Number of Anti-retroviral Medications Taken in Combination With Tipranavir/Ritonavir
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Number; unit: participants
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
participants
  < 6 | 30
  6 - 10 | 15
  11 - 15 | 16
  > 15 | 3
  missing | 1

10. Secondary Outcome: Use of Lipid Lowering Agents During the Study
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Number; unit: participants
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
participants
  No | 59
  Yes | 6

11. Secondary Outcome: Body Mass Index Class (Kilograms/Square Meter)
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Number; unit: participants
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
participants
  Low (< 18) | 2
  Normal (18 - 30) | 62
  High (> 30) | 0
  missing | 1

12. Secondary Outcome: Total Cholesterol Over Time
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
mg/dl
  Month 1 (n=42) | 213.0 [179.0 to 233.0]
  Month 3 (n=41) | 214.0 [175.0 to 229.0]
  Month 6 (n=48) | 213.0 [189.3 to 240.0]
  Month 9 (n=37) | 217.0 [177.0 to 235.0]
  Month 12 (n=35) | 216.0 [177.9 to 232.0]

13. Secondary Outcome: High Density Lipoprotein (HDL) Cholesterol Over Time
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
mg/dl
  Month 1 (n=28) | 38.0 [35.5 to 47.0]
  Month 3 (n=29) | 39.0 [35.0 to 45.0]
  Month 6 (n=32) | 39.5 [34.6 to 47.0]
  Month 9 (n=28) | 39.0 [33.5 to 48.0]
  Month 12 (n=27) | 37.0 [33.0 to 53.0]

14. Secondary Outcome: Low Density Lipoprotein (HDL) Cholesterol Over Time
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
mg/dl
  Month 1 (n=23) | 120.0 [88.0 to 147.0]
  Month 3 (n=25) | 123.0 [99.0 to 134.0]
  Month 6 (n=29) | 125.0 [110.0 to 147.0]
  Month 9 (n=26) | 117.5 [98.0 to 132.0]
  Month 12 (n=23) | 122.0 [102.0 to 138.0]

15. Secondary Outcome: Triglycerides Over Time
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
mg/dl
  Month 1 (n=38) | 237.5 [143.0 to 479.0]
  Month 3 (n=39) | 256.9 [160.0 to 361.0]
  Month 6 (n=46) | 246.0 [190.0 to 361.0]
  Month 9 (n=33) | 283.4 [186.0 to 330.0]
  Month 12 (n=32) | 265.5 [171.0 to 458.5]

16. Secondary Outcome: Alanine Aminotransferase (ALT) Over Time
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Median (Inter-Quartile Range); unit: international units/liter
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
international units/liter
  Month 1 (n=52) | 33.0 [25.7 to 48.5]
  Month 3 (n=49) | 31.0 [24.0 to 50.0]
  Month 6 (n=55) | 37.0 [27.0 to 51.0]
  Month 9 (n=41) | 34.0 [28.0 to 53.0]
  Month 12 (n=42) | 37.5 [29.0 to 54.0]

17. Secondary Outcome: Aspartate Aminotransferase (ALT) Over Time
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Median (Inter-Quartile Range); unit: international units/liter
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
international units/liter
  Month 1 (n=54) | 34.5 [25.0 to 55.0]
  Month 3 (n=50) | 33.5 [23.0 to 55.0]
  Month 6 (n=57) | 40.0 [25.0 to 62.0]
  Month 9 (n=44) | 44.0 [27.0 to 62.0]
  Month 12 (n=42) | 37.5 [29.0 to 53.0]

18. Secondary Outcome: Gamma-glutamyl Transpeptidase (GGT) Over Time
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Median (Inter-Quartile Range); unit: international units/liter
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
international units/liter
  Month 1 (n=54) | 72.0 [41.0 to 121.0]
  Month 3 (n=49) | 72.0 [50.0 to 164.0]
  Month 6 (n=57) | 72.0 [56.0 to 154.0]
  Month 9 (n=44) | 76.0 [48.0 to 128.0]
  Month 12 (n=43) | 68.0 [50.0 to 104.0]

19. Secondary Outcome: Creatinine Over Time
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
mg/dl
  Month 1 (n=43) | 0.90 [0.80 to 1.00]
  Month 3 (n=46) | 0.90 [0.80 to 1.01]
  Month 6 (n=49) | 0.90 [0.80 to 1.00]
  Month 9 (n=35) | 0.90 [0.80 to 1.07]
  Month 12 (n=33) | 0.90 [0.80 to 1.00]

20. Secondary Outcome: Total Bilirubin Over Time
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
mg/dl
  Month 1 (n=39) | 0.42 [0.34 to 0.60]
  Month 3 (n=38) | 0.40 [0.33 to 0.60]
  Month 6 (n=43) | 0.50 [0.38 to 0.60]
  Month 9 (n=31) | 0.50 [0.40 to 0.60]
  Month 12 (n=32) | 0.40 [0.36 to 0.51]

21. Secondary Outcome: Alkaline Phosphatase Over Time
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), all patients entered and treated
Measure: Median (Inter-Quartile Range); unit: international units/liter
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Number analyzed (Participants) | 65
international units/liter
  Month 1 (n=33) | 90.0 [76.0 to 111.0]
  Month 3 (n=38) | 92.5 [76.0 to 103.5]
  Month 6 (n=26) | 87.5 [80.0 to 114.0]
  Month 9 (n=24) | 86.5 [79.0 to 118.0]
  Month 12 (n=43) | 92.5 [76.2 to 108.5]

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Aptivus® in Combination With Low-dose Norvir®
Serious Adverse Events (participants affected / at risk) | 3/65
Other Adverse Events (participants affected / at risk) | 4/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aptivus® in Combination With Low-dose Norvir® (N=65)
Death (General disorders) | 1
Transaminases increased (Investigations) | 1
Pulmonary embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aptivus® in Combination With Low-dose Norvir® (N=65)
Nausea (Gastrointestinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.